CLINICAL TRIAL: NCT03010007
Title: Prospective Analysis of Seasonal Influenza - Viral Transmission and Evolution in the City of Basel, Switzerland [Prospektive Systemanalyse Der Saisonalen Influenza - Virustransmission Und Evolution in Der Stadt Basel] in German
Brief Title: Prospective Analysis of Seasonal Influenza - Viral Transmission and Evolution in the City of Basel, Switzerland
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Swiss Federal Institute of Technology (Other); University Children's Hospital Basel (Other); University of Basel (Other)
Responsible Party: Sponsor
Other Study IDs: Influenza in Basel 2016/2017
Record Dates: First submitted 2016-12-22; First posted 2017-01-04 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Influenza
Keywords: Influenza; High-Throughput Nucleotide Sequencing; Viral Transmission
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood (serum) and nasopharyngeal swabs
Oversight: Data Monitoring Committee: No

SUMMARY:
Influenza associated illness has a global annual impact with high morbidity and mortality. Transmission mechanisms and rates are under-investigated and overall poorly understood.

This project aims to use epidemiological tools to understand the transmission and evolution of influenza viruses at an individual and population level within a small-scale city (Basel) through a combination of experimental, clinical and mathematical advances. The investigators aim to quantitatively characterize the viral transmission using novel molecular-epidemiological tools based on whole genome sequencing.

DETAILED DESCRIPTION:
In this prospective observational study, paediatric and adult outpatients presenting with influenza-like illness will be enrolled at the emergency departments of the University Hospital Basel (USB), the paediatric University Hospital of both Basel (UKBB), or a network of family doctors (associated with Center of Primary Health Care).

The Clinical Trial Unit at the University Hospital Basel will coordinated the recruitment process, collect data and sample all patients during the influenza season 2016/17. Samples will be collected such as whole blood, serum and DNA, nasopharyngeal swamps to diagnose influenza by polymerase chain reaction (PCR) assay and to determine colonization rates with Staphylococcus aureus and Streptococcus pneumonia. All samples except the first naso-pharyngeal swab for influenza diagnostics will be stored in a biobank and analysed in batches. Each influenza virus isolate will be sequenced using a "whole genome sequencing" approach. The viral transmission and evolution will be analysed using whole genome data for a detailed molecular and phylogenetic tree analysis, respectively. The epidemiological and geographical data will be incorporated into the phylogenetic model.

Specific aims are:

(i) to determine the impact of the most important epidemiological parameters, first focusing on the age profile, followed by children per house hold, and population density, on influenza transmission at an individual and population level, drawing on an analysis of baseline humoral immunity and whole genome sequencing data, (ii) to understand the viral evolution during seasonal epidemics, (iii) to develop dynamic mathematical models that are able to predict viral transmission and evolution based on the retrospective results from (i) and (ii) and to validate this model in future influenza seasons.

To realize the interdisciplinary approach, the investigators will rely on the expertise in mathematical modelling of viral epidemiology and evolution and established geographical expertise, next generation sequencing, clinical epidemiology, and immunologic diagnostic techniques.

ELIGIBILITY:
Inclusion Criteria:

* Each pediatric or adult patient, which fulfill the Worl Health Organization (WHO) definition of Influenza like illness.
* The case definition includes an acute respiratory infection with coughing, fever ≥38°C, and start of symptoms within the last 10 days.
* Presentation of the patient with influenza-like illness on the emergency ward of the University Hospital Basel or the University Children Hospital of both Basel or a collaborating private practise.
* Patient has to live in the city of Basel.

Exclusion Criteria:

* Patients who are not living in the City of Basel.
* Case definition for influenza like illness is not fulfilled.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Paediatric or adult patients fulfilling the World Health Organization (WHO) definition of an influenza-like illness. A total number of 1000 influenza PCR-confirmed cases should be included.
Sampling Method: Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2017-01; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Investigation of the phylogenetic relation of viral isolates from participating patients using whole-genome sequencing and bioinformatics | Baseline
  The primary microbiological endpoint is the connection of two viral isolates via comparison and phylogenetic analysis by using the genetic information

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Egli, PD Dr. FAMH, Principal Investigator — Clinical Microbiology, University Hospital Basel
Locations (4):
- Switzerland (4):
  - Federal Institute of Technology Zurich, Basel
  - University Children's Hospital, Basel
  - University Hospital Basel, Basel
  - Universitätres Zentrum für Hausarztmedizin beider Basel, University of Basel, Basel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Egli A, Saalfrank C, Goldman N, Brunner M, Hollenstein Y, Vogel T, Augustin N, Wuthrich D, Seth-Smith HMB, Roth E, Syedbasha M, Mueller NF, Vogt D, Bauer J, Amar-Sliwa N, Meinel DM, Dubuis O, Naegele M, Tschudin-Sutter S, Buser A, Nickel CH, Zeller A, Ritz N, Battegay M, Stadler T, Schneider-Sliwa R. Identification of influenza urban transmission patterns by geographical, epidemiological and whole genome sequencing data: protocol for an observational study. BMJ Open. 2019 Aug 20;9(8):e030913. doi: 10.1136/bmjopen-2019-030913. PMID 31434783